CLINICAL TRIAL: NCT02788344
Title: Baseline Characteristics, Processes of Care, System-related Factors, and Clinical Outcomes Associated With the Quality and Safety of Initial Management for ST-segment Elevation Myocardial Infarction: A Multicenter Cohort Study
Brief Title: Quality and Safety of Initial Management for ST-segment Elevation Myocardial Infarction
Acronym: STEMI-Qual
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: PREPS14-0040
Record Dates: First submitted 2016-05-18; First posted 2016-06-02 (Estimated); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Infarction
Keywords: Observational study; Myocardial revascularization; Thrombolytic therapy; Hospital mortality; Hemorrhage; Quality of health care; Angioplasty
MeSH Terms: conditions — Myocardial Infarction; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Daily practice care for patients with suspected of STEMI — N/A: Practice care evaluation in real-life setting

SUMMARY:
This is a multicenter multidisciplinary study designed to investigate patient, provider, and system-related factors that are associated with the quality and safety of initial management for suspected ST-segment elevation myocardial infarction (STEMI) evolving for less than 12 hours in daily practice. The primary hypotheses are that delayed reperfusion therapy for suspected STEMI independently relates to provider practice patterns and system barriers. It is further postulated that non-compliance with target delays in implementing percutaneous coronary intervention (PCI) or fibrinolytic therapy is associated with worse in-hospital clinical outcomes. The secondary hypotheses are that the delivery of acute reperfusion therapy within target delays is associated with increased rates of false-positive cardiac catheterization laboratory activation, inadvertent fibrinolytic therapy, and bleeding events.

The project will be conducted in three emergency medical services and 23 public and private (for-profit and non-for-profit) acute care hospitals in Northern Alps in France. Data over the index hospital stay period will be retrospectively collected for all the patients included in an ongoing prospective regional hospital-based clinical registry of suspected STEMI from October, 1st, 2002 to December, 31, 2014. Inclusion of 7435 patients is anticipated.

In this observational retrospective study, no specific intervention is assigned to participants. All diagnostic testing, procedures, and medication ordering are performed at the discretion of attending physicians. No enrollment or follow-up visits are planned.

The primary effectiveness outcome is timely acute reperfusion therapy. The secondary effectiveness outcomes include false-positive cardiac catheterization laboratory activation for catheterization candidates and inadvertent fibrinolytic therapy. The secondary medical outcomes include in-hospital all-cause mortality, major adverse cardiovascular events, and major bleeding events. Multivariable logistic regression model will be developed to identify baseline characteristics that are independently associated with timely acute reperfusion therapy. Propensity score analysis will be performed for comparing clinical outcomes between timely acute reperfusion therapy recipients and non-recipients.

DETAILED DESCRIPTION:
Objectives

The broad objectives of this multicenter and multidisciplinary observational cohort study are to investigate patient, provider, and system-related factors that are associated with the quality and safety of initial management for suspected ST-segment elevation myocardial infarction (STEMI) evolving for less than 12 hours in daily practice. The findings of this study should help identifying areas with room for improvement in clinical pathway for STEMI patients. The specific aims of this project are:

* to investigate the independent associations between the delivery of timely acute reperfusion therapy and patient, provider, and system-related factors, according to current guidelines
* to assess the independent associations between the delivery of timely acute reperfusion therapy and in-hospital clinical outcomes (including all-cause mortality and major adverse cardiovascular events)
* to determine the independent risk factors for major bleeding (excluding coronary-artery bypass graft-related bleeding events) among baseline patient and provider characteristics, processes of care, and system-related factors, respectively
* to elucidate the prevalence, risk factors, and in-hospital clinical outcomes independently associated with false-positive cardiac catheterization laboratory activation or inadvertent fibrinolytic therapy
* to determine how hospitals are interconnected by transferring patients with suspected STEMI

Hypotheses The primary hypotheses guiding this project are that delayed reperfusion therapy for suspected STEMI independently relates to provider practice patterns and system barriers. It is further postulated that non-compliance with target delays in implementing primary PCI or fibrinolytic therapy is associated with worse in-hospital clinical outcomes.

The secondary hypotheses are that the delivery of acute reperfusion therapy within target delays is associated with increased rates of false-positive cardiac catheterization laboratory activation, inadvertent fibrinolytic therapy, and bleeding events.

Participating study centers and setting The project will be conducted at 3 emergency medical services (EMS/SAMU) and 23 public and private (for-profit and non-for-profit) acute care hospitals in Northern Alps in France. Northern Alps are a predominantly mountainous area covering 15,000 km² with an estimated population of 1,860,000 inhabitants with large seasonal variations due to tourism. The median distance and driving time from each community hospital to the closest PCI center are 63 km (range, 4.5-132 km) and 43 min (range, 10-88 min), respectively.

As part of a coordinated regional system of reperfusion therapy for STEMI, all participating centers have a long collaborative tradition in STEMI management research.The rationale, data collection methods, verification procedures, and primary outcomes of this registry have been reported in detail elsewhere.

Baseline data collection methods

1. Prospective data collection As part of the ongoing registry, attending physicians or clinical research technicians routinely abstract summary information on demographics, presenting characteristics (including electrocardiographic findings), coronary angiography findings, and delivery and timing of acute reperfusion therapy in both prehospital and hospital settings.

   Based on patient home address, travel time and travel distance to the nearest community hospital and PCI-capable hospital will be obtained through calls to commercial Web page (MapQuest or Via Michelin). ZIP code will replace patient home address when unavailable. Previous studies have shown that this method provides reasonable estimates. To account for peak travel time, slowdowns of 20% will be factored in during the hours of 7 to 9 AM and 4 to 7 PM, Monday through Friday.
2. Retrospective data collection Two clinical research nurses will perform retrospective chart review using a computerized data collection instrument. The following variables will be recorded: baseline patient characteristics, clinical variables, comorbid conditions, laboratory variables, procedural interventions (cardiac catheterization, PCI [not primary], and coronary artery bypass grafting) at any time during index hospitalization, medications (on admission, during the first 24 hours, and at discharge). Index hospitalization includes both admitting and transfer hospital stays.

Characteristics will also be collected for attending physicians (gender, age, discipline) as well as admitting and transfer hospitals (community vs PCI-capable facility, size, public or non for profit versus for profit). Consistent with a previous study, PCI centers are defined as hospitals that offer emergency PCI 24 h a day, 7 days a week.

Data management

1. Prospective data collection As part of the ongoing registry, data are prospectively recorded in duplicate on standardized forms designed to facilitate data collection and entry. All completed forms are forwarded to the core coordinating facility of the regional emergency system (RENAU=Réseau Nord-Alpin des Urgences ; www.renau.org), where the data are entered electronically (single-data entry) and maintained on a local computer network. The data entry screens are similar to the paper forms. Original data collection forms are kept in locked file cabinets.

   Data integrity is enforced through two complementary approaches:
   * Routine edit checks (valid values, range checks, and consistency checks) are performed at the time of data entry by a clinical research technician at the core coordinating facility.
   * The registry statistician periodically screens data for additional errors using programs designed to detect missing values or inconsistencies.
2. Retrospective data collection To ensure optimal quality, all data collected retrospectively by chart review will be entered electronically by clinical research nurses using a personal identification code and password-protected web-based data collection system. The clinical research nurses will receive formal training in the methods of data abstraction and recording. An operation manual that includes definitions and acceptable data sources for all variables will be distributed. Reliability of data abstraction will be assessed by randomly selecting 30 cases for independent collection by the two study nurses.

The data manager will screen data for additional errors using programs designed to detect missing values or inconsistencies.

Statistical analysis

1. Overview Standard descriptive summary statistics will be used for reporting continuous and categorical variables. In univariate analysis, inferential comparisons will be performed using analysis of variance or the Kruskal-Wallis rank sum test. Logarithm transformation may be used for highly skewed variables prior to inferential comparisons. Categorical variables will be analyzed with the use of Khi² or Fisher exact tests. Trends across ordered groups will be analyzed for statistical significance using the Khi² test for trends for categorical variables and the non-parametric Wilcoxon-type test for trends for continuous variables, respectively. Two-sided P values of less than 0.05 will be considered statistically significant.
2. Primary effectiveness outcome A non-parsimonious multivariable logistic regression model will be developed to identify baseline characteristics that are independently associated with timely acute reperfusion therapy. Covariates entered into the multivariable model will be prespecified before modelling, without investigating their association with the primary study outcome.

   Secondary analysis restricted to the subset of patients with prehospital management will use multilevel logistic regression, with the 3 levels defined by patients, mobile intensive care units, and hospitals. The Metropolis-Hastings algorithm (a Markov Chain Monte Carlo method) will be used to account for the cross-classification of mobile intensive care units that transported patients at more than one study site.
3. Secondary medical outcomes Because timely acute reperfusion therapy is not randomly assigned in this observational study, unadjusted comparisons of medical outcomes between study groups might be confounded by imbalances in baseline characteristics.For this purpose, propensity score analysis that compensate for differences in measured baseline characteristics will be performed between timely acute reperfusion therapy recipients and non-recipients.

   Practically, a propensity score will be derived for the receipt of timely acute reperfusion therapy using a full non-parsimonious logistic regression model that includes baseline characteristics as covariates.

   Each patient will be assigned a propensity score, which may range from 0.00 to 1.00 and reflects the conditional probability of timely acute reperfusion receipt given his baseline characteristics.

   To compare secondary medical outcomes among patients with similar conditional probability of timely acute reperfusion therapy, a cohort of timely acute reperfusion therapy recipients and non-recipients matched by propensity score will be also defined. For this purpose, an algorithm will be used to match each timely acute reperfusion therapy recipient to a single non-recipient who have the nearest propensity score within one digit. If this cannot not be done, that timely acute reperfusion therapy recipient will be excluded from the propensity-matched analysis. The propensity-matched cohort will be evaluated for significant residual imbalances in baseline characteristics. Then logistic regression will be used to estimate the odds ratio for each secondary medical outcomes associated with the receipt of timely acute reperfusion therapy among propensity score-matched patients.
4. Secondary effectiveness outcomes Using the same modelling approach as previously described (i.e., b. primary effectiveness outcome), multivariable logistic regression will be performed to identify baseline characteristics that are independently associated with false-positive cardiac catheterization laboratory activation among patients who are candidate for primary PCI. A first-order interaction term involving prehospital cardiac catheterization laboratory activation will be tested for statistical significance. If appropriate, analysis will be stratified according to prehospital versus hospital cardiac catheterization laboratory activation. Then medical outcomes will be compared between false positive and true positive cardiac catheterization laboratory activation after adjusting for quintile of propensity score.

In a separate analysis, multivariate logistic regression will be performed to identify baseline characteristics that are independently associated with inadvertent fibrinolytic therapy among fibrinolysis recipients. A first-order interaction term involving prehospital fibrinolysis will be tested for statistical significance and, if appropriate, analysis will be stratified according to the receipt of prehospital versus hospital fibrinolysis. Then odds ratio will be estimated for each medical outcome associated with inadvertent fibrinolysis after adjusting for quintile of propensity score.

Harms and safety In this retrospective observational study, severe adverse events occurring during hospitalization will be specified as secondary medical study outcomes (mortality, major adverse cardiac events [reinfarction, cardiogenic shock, cardiac arrest, heart failure, stroke], and major bleeding).

Other prespecified adverse events will be recorded, including atrial fibrillation or flutter, sustained ventricular tachycardia, atrioventricular block (Mobitz II or 3rd degree), mechanical complications (ventricular septal defect, mitral regurgitation, free wall rupture), venous thromboembolism (deep vein thrombosis and/or pulmonary embolism), acute renal failure, thrombocytopenia and heparin-induced thrombocytopenia, and non-major bleeding events.

Adverse events will be collected through a structured chart review. There will be no attempt to determine potential causality.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older
* who are alive at first medical contact
* with symptoms suggestive of myocardial infarction (chest pain lasting for more than 20 minutes and not responsive to nitrates),
* occuring between October, 1st, 2002 and December, 31, 2014
* evolving for less than 12 hours from symptom onset,
* and with evidence of persistent ST-segment elevation of at least 1 mm in two or more limb leads, ST-segment elevation of at least 2 mm in two or more precordial leads, or new or presumed new left bundle branch block.

Exclusion Criteria:

* patients who refused the use of their medical data
* patient already hospitalized when STEMI occured, whatever the reason of hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older with symptoms suggestive of myocardial infarction (chest pain lasting for more than 20 minutes and not responsive to nitrates).
  Eligible patients are enrolled irrespective of final discharge diagnosis of STEMI, other acute coronary syndrome (non-ST-segment elevation myocardial infarction, unstable angina pectoris), other cardiac disease, or non-cardiac disease.
Sampling Method: Probability Sample
Enrollment: 6920 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Fibrinolytic therapy within 30 minutes of first medical contact | 30 minutes
primary PCI within 60 minutes for early presenters or patients, presenting directly to a PCI capable hospital | 60 minutes
primary PCI within 90 minutes of first medical contact for all patients | 90 minutes

SECONDARY OUTCOMES:
In-hospital all-cause mortality | up to 2 weeks, from the day of myocardial infarction's onset to the first hospital discharge
  patients are hospitalized the day of myocardial infarction's onset, and usually discharged from hospital a few days later. It is possible that this time frame was shortened between 2002 and 2014
In-hospital major adverse cardiovascular events (reinfarction, cardiogenic shock, heat failure, stroke, cardiac arrest) | up to 2 weeks, from the day of myocardial infarction's onset to the first hospital discharge
  patients are hospitalized the day of myocardial infarction's onset, and usually discharged from hospital a few days later. It is possible that this time frame was shortened between 2002 and 2014
In-hospital major bleeding events | up to 2 weeks, from the day of myocardial infarction's onset to the first hospital discharge
  patients are hospitalized the day of myocardial infarction's onset, and usually discharged from hospital a few days later. It is possible that this time frame was shortened between 2002 and 2014

CONTACTS AND LOCATIONS:
Overall Officials: Loïc E BELLE, MD, Study Chair — CH Annecy Genevois, head of RENAU (Réseau Nord Alpin des Urgences); José LABARERE, MD, PhD, Study Chair — Centre Hospitalier Universitaire Grenoble Alpes, France; Gérald VANZETTO, MD, PhD, Study Chair — Centre Hospitalier Universitaire Grenoble Alpes, France
Locations (1):
- RENAU network, Metz-Tessy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Belle L, Fourny M, Reynaud T, Hammer L, Vanzetto G, Labarere J; RENAU-RESURCOR study investigators. Efficacy and safety of glycoprotein IIb/IIIa receptor antagonists for patients undergoing percutaneous coronary intervention within twelve hours of fibrinolysis. Catheter Cardiovasc Interv. 2011 Sep 1;78(3):376-84. doi: 10.1002/ccd.22825. Epub 2011 Mar 16. PMID 21413113
- [Background] Belle L, Labarere J, Fourny M, Drouet E, Mulak G, Dujardin JJ, Vilarem D, Bonnet P, Hanssen M, Simon T, Ferrieres J, Danchin N; French registry of Acute ST elevation or non-ST-elevation Myocardial Infarction study investigators. Quality of care for myocardial infarction at academic and nonacademic hospitals. Am J Med. 2012 Apr;125(4):365-73. doi: 10.1016/j.amjmed.2011.11.015. PMID 22444102
- [Background] Belle L, Motreff P, Mangin L, Range G, Marcaggi X, Marie A, Ferrier N, Dubreuil O, Zemour G, Souteyrand G, Caussin C, Amabile N, Isaaz K, Dauphin R, Koning R, Robin C, Faurie B, Bonello L, Champin S, Delhaye C, Cuilleret F, Mewton N, Genty C, Viallon M, Bosson JL, Croisille P; MIMI Investigators*. Comparison of Immediate With Delayed Stenting Using the Minimalist Immediate Mechanical Intervention Approach in Acute ST-Segment-Elevation Myocardial Infarction: The MIMI Study. Circ Cardiovasc Interv. 2016 Mar;9(3):e003388. doi: 10.1161/CIRCINTERVENTIONS.115.003388. PMID 26957418
- [Background] Beygui F, Cayla G, Roule V, Roubille F, Delarche N, Silvain J, Van Belle E, Belle L, Galinier M, Motreff P, Cornillet L, Collet JP, Furber A, Goldstein P, Ecollan P, Legallois D, Lebon A, Rousseau H, Machecourt J, Zannad F, Vicaut E, Montalescot G; ALBATROSS Investigators. Early Aldosterone Blockade in Acute Myocardial Infarction: The ALBATROSS Randomized Clinical Trial. J Am Coll Cardiol. 2016 Apr 26;67(16):1917-27. doi: 10.1016/j.jacc.2016.02.033. PMID 27102506
- [Background] Fourny M, Lucas AS, Belle L, Debaty G, Casez P, Bouvaist H, Francois P, Vanzetto G, Labarere J. Inappropriate dispatcher decision for emergency medical service users with acute myocardial infarction. Am J Emerg Med. 2011 Jan;29(1):37-42. doi: 10.1016/j.ajem.2009.07.008. Epub 2010 Mar 9. PMID 20825772
- [Background] Labarere J, Belle L, Fourny M, Vanzetto G, Debaty G, Delgado D, Brallet J, Vallet B, Danchin N; USIC 2000; FAST-MI. Regional system of care for ST-segment elevation myocardial infarction in the Northern Alps: a controlled pre- and postintervention study. Arch Cardiovasc Dis. 2012 Aug-Sep;105(8-9):414-23. doi: 10.1016/j.acvd.2012.05.001. Epub 2012 Jul 17. PMID 22958884
- [Background] Labarere J, Belle L, Fourny M, Genes N, Lablanche JM, Blanchard D, Cambou JP, Danchin N; Unite de Soins Intendifs Coronaires 2000 Inverstigators. Outcomes of myocardial infarction in hospitals with percutaneous coronary intervention facilities. Arch Intern Med. 2007 May 14;167(9):913-20. doi: 10.1001/archinte.167.9.913. PMID 17502532
- [Background] Raskovalova T, Twerenbold R, Collinson PO, Keller T, Bouvaist H, Folli C, Giavarina D, Lotze U, Eggers KM, Dupuy AM, Chenevier-Gobeaux C, Meune C, Maisel A, Mueller C, Labarere J. Diagnostic accuracy of combined cardiac troponin and copeptin assessment for early rule-out of myocardial infarction: a systematic review and meta-analysis. Eur Heart J Acute Cardiovasc Care. 2014 Mar;3(1):18-27. doi: 10.1177/2048872613514015. Epub 2013 Nov 20. PMID 24562800
- [Background] Yayehd K, Ricard C, Ageron FX, Buscaglia L, Savary D, Audema B, Lacroix D, Barthes M, Joubert P, Gheno G, Belle L; RENAU-RESURCOR study investigators. Role of primary care physicians in treating patients with ST-segment elevation myocardial infarction located in remote areas (from the REseau Nord-Alpin des Urgences [RENAU], Network). Eur Heart J Acute Cardiovasc Care. 2015 Feb;4(1):41-50. doi: 10.1177/2048872614544856. Epub 2014 Jul 29. PMID 25075005